CLINICAL TRIAL: NCT03625102
Title: A Randomized, Double-Blind, Dosing-Ranging, Placebo-controlled Trial of Antroquinonol in Patients With Chronic Hepatitis B
Brief Title: A Randomized, Double-Blind Trial of Antroquinonol in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Golden Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GHHBV-2-001
Record Dates: First submitted 2018-08-05; First posted 2018-08-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: HBV
Keywords: Antroquinonol; Hocena
MeSH Terms: interventions — antroquinonol

STUDY DESIGN:
Intervention Model Description: This is a single-center, phase IIa, double blind, and randomized, placebo-controlled trial of Antroquinonol in patients with hepatitis B infection. Subjects with diagnosis of hepatitis B meet inclusion/exclusion criteria will be randomized into 3 groups:
  1. Antroquinonol 100 mg PO BID
  2. Antroquinonol 50 mg PO BID
  3. Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antroquinonol 100 mg PO BID (Experimental): Antroquinonol (Hocena) 50mg/capsule. 2 capsules antroquinonol, twice a day.
  Interventions: Drug: Antroquinonol
- Antroquinonol 50 mg PO BID (Experimental): Antroquinonol (Hocena) 50mg/capsule. 1 capsule antroquinonol and 1 capsule placebo,twice a day.
  Interventions: Drug: Antroquinonol; Other: placebo
- Placebo (Placebo Comparator): Placebo capsule, 2 capsules placebo, twice a day
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Antroquinonol — Antroquinonol will be provided as a capsule-shaped which contain 50 mg Antroquinonol.
  Other Names: Hocena
  Arms: Antroquinonol 100 mg PO BID; Antroquinonol 50 mg PO BID
Other: placebo — The matching placebo will be packaged as Antroquinonol with appearance identical in all aspects
  Arms: Antroquinonol 50 mg PO BID; Placebo

SUMMARY:
Hepatitis B virus infection is a worldwide disease and is still the most common cause of hepatocellular carcinoma (HCC).Existing treatments for hepatitis B infection have various side-effects including renal toxicity and drug resistance or failure.

DETAILED DESCRIPTION:
Hepatitis B virus infection is a worldwide disease and is still the most common cause of hepatocellular carcinoma (HCC). Those carriers in China account for 33% of all chronic carriers globally. A big epidemiological study of patients with chronic hepatitis B has revealed that baseline HBV DNA level or cirrhosis is an independent predictor for the occurrence of HCC.

Antroquinonol is a new chemical entity isolated from the mycelium of Antrodia camphorata, which showed interesting anticancer and anti-inflammatory activities.Previous studies have indicated that signaling molecules, such as PI3K, AMPK, and mTOR, participate in Antroquinonol-induced cancer cell death, whereas Nrf2 and NF-kB are involved in the anti-inflammatory effects of Antroquinonol. Moreover, we also found the administration of Antroquinonol also differentially modulated T cell activity and reduced IL-18 production, but enhanced the activation of Nrf2 and, thus, suppressed oxidative stress by animal studies. These results demonstrate the potential applications of Antroquinonol in treating hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HBV infection patients between the ages of 20 and 75 years with serum hepatitis B surface antigen(HBsAg) positivity for more than 6 months
2. BMI≦35
3. HBsAg≧10 IU/mL and HBV DNA≧2000 IU/mL.
4. AST or ALT≧25 IU and ALT<5xULN
5. Female subject must use effective methods of contraception.
6. No abnormal finding of clinical relevance
7. Written informed consent

Exclusion Criteria:

1. Evidence of hepatic decompensation such as:

   1. Coagulopathy defined as prolongation of prothrombin time greater than 3 seconds
   2. Total bilirubin of 2 times the upper limit of normal
   3. FIB-4 of 3.25 or greater
2. Abnormal hematological and biochemical parameters at screening A、 White blood cell count less than 2500 cells/uL B、 Absolute neutrophil count (ANC) less than 1,000 cells/mm3 (less than 750 mm3 for African or African-American subjects) C、 Hemoglobin less than 12 g/dL for males, less than 11 g/dL for females D、 Estimated GFR less than 50 mL/min
3. Suspected or confirmed liver diseases from etiologies other than HBV (such as alcohol, toxin, drug, shock, acute viral hepatitis A or E), co-infection with human immunodeficiency virus, hepatitis C virus or hepatitis delta virus, prior antiviral treatment with NUCs or interferon, and recent immunosuppressive therapy (including chemotherapy and systemic corticosteroid).
4. Immunodeficiency disorders or severe autoimmune disease
5. Severe pulmonary disorders or significant cardiac diseases
6. Gastrointestinal disorder with post-operative condition that could interfere with drug absorption
7. Significant psychiatric illness that in the judgment of the Investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent
8. Any malignancy diagnosed within 5 years or evidence of hepatocellular carcinoma (e.g., α fetoprotein > 50ng/mL or radiologic evidence)
9. Solid organ transplantation
10. Current drug or alcohol abuse
11. Pregnancy or lactation
12. Under hepatitis B antiviral or interferon treatment within 3 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Percentage | 12 weeks
  The percentage improvement between baseline and day 85 in quantitative HBsAg.

SECONDARY OUTCOMES:
IU/mL | 4 week
  Sserum hapatitis B virus DNA level
score | 12 week
  The Fibrosis-4 score helps to estimate the amount of scarring in the liver
Unit/L | 4 week
  Glutamic Oxaloacetic Transaminase
Unit /L | 4 week
  Glutamic Pyruvic Transaminase

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Pin Lin, MD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No